CLINICAL TRIAL: NCT02712307
Title: A Randomized Controlled Study of 5 and 10 Days Treatment With Phenoxymethylpenicillin for Pharyngotonsillitis Caused by Streptococcus Group A
Brief Title: Study of 5 and 10 Days Treatment With Penicillin Against Sore Throat Caused by Streptococci
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ass. Prof. Katarina Hedin (Other Government)
Responsible Party: Sponsor-Investigator, Ass. Prof. Katarina Hedin, Professor, Public Health Agency of Sweden
Organization: Public Health Agency of Sweden (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoHM/Tonsillit2015; 2015-001752-30 (EudraCT Number)
Record Dates: First submitted 2016-03-04; First posted 2016-03-18 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Penicillin V

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 days (Experimental): Phenoxymethylpenicillin 800 mg x 4 for 5 days
  Interventions: Drug: Phenoxymethylpenicillin
- 10 days (Active Comparator): Phenoxymethylpenicillin 1000 mg x 3 for 10 days
  Interventions: Drug: Phenoxymethylpenicillin

INTERVENTIONS:
Drug: Phenoxymethylpenicillin
  Other Names: Penicillin V

SUMMARY:
The primary objective of the study is to compare the clinical efficacy of 5 days (800 mg x 4) versus 10 days (1000 mg x 3) treatment with phenoxymethylpenicillin (PcV) in adults, adolescents and children with streptococcal tonsillitis. Patients are recruited from 17 primary Health care centres in the south of Sweden. Adult men and women, youth and children ≥ 6 years of age who are visiting the primary Health care for sore throat with suspected tonsillitis and meeting the criteria in accordance with current treatment recommendations for pharyngotonsillitis, ie 3-4 Centor criteria (fever≥ 38.5, tender lymph nodes, coatings of the tonsils and absence of cough) and a positive rapid antigen detection test (RADT) for Group A streptococcus (GAS) will be included in the study. Patients will be randomized to be prescribed PcV of 5 and 10 days. Each patient or guardian fills daily in a short diary including aches, fever, PcV doses, pain relievers, adverse events etc. Five to seven days after last intake of PcV the general practioner make a clinical judgement if the patient has recovered from the pharyngotonsillitis. Questions to be asked are if remaining symptoms or new symptoms of sore throat is present, if adverse events have been noted or of any extra physician visits have been made. Throat swab for semi quantitative cultures of Streptococcus group A, C and G are made at randomization and five to seven days after last intake of PcV. A study nurse will contact the patients one month and three months after the last treatment day for follow-up. If the patient has reconsulted or been hospitalised for a sore throat or possible complication, those patient records will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Adults, adolescents and children ≥ 6 years of age with verified streptococcal pharyngotonsillitis.

Exclusion Criteria:

* Signs of serious infection.
* Known hypersensitivity against penicillin.
* Chronic disease with effect on the immune response.
* Immunosuppressive treatment.
* Streptococcal tonsillitis within one month (relapse).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Clinical cure | 5-7 days after discontinuation of treatment
  Difference between treatment groups in the rate of clinical cure. Clinical cure is defined as clinical judgement by physician and absence of Centor criteria (coating, fever and swollen Large Granular Lymphocyte glands).

SECONDARY OUTCOMES:
Bacteriological cure | 5-7 days after discontinuation of treatment
  Difference between treatment groups in the rate of bacteriological cure, defined as absence of GAS in culture.
Frequency of relapses | 1 month after discontinuation of treatment
Frequency of complications | Within 3 months after discontinuation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sigvard Mölstad, Professor, Principal Investigator — Lund University; Katarina Hedin, MD PhD, Principal Investigator — Department of Research and Development, Region Kronoberg and Lund University; Pär-Daniel Sundvall, MD PhD, Principal Investigator — Research and Development Unit, Primary Health Care in Southern Älvsborg County and University of Gothenburg
Locations (17):
- Sweden (17):
  - Alvesta vårdcentral, Alvesta
  - Närhälsan Bollebygd vårdcentral, Bollebygd
  - Capio Citykliniken Bunkeflo Hyllie, Bunkeflostrand
  - Vårdcentralen Tåbelund, Eslöv
  - Närhälsan Fristad vårdcentral, Fristad
  - Vårdcentralen Lessebo, Lessebo
  - Capio Citykliniken Malmö Limhamn, Limhamn
  - Löddeköpinge vårdcentral, Löddeköpinge
  - Vårdcentralen Sorgenfrimottagningen, Malmo
  - Vårdcentralen Lundbergsgatan, Malmo
  - Närhälsan Sandared vårdcentral, Sandared
  - Vårdcentrlaen Sjöbo, Sjöbo
  - Närhälsan Billingen vårdcentral, Skövde
  - Närhälsan Norrmalm vårdcentral, Skövde
  - Närhälsan Södra Ryd, Skövde
  - Vårdcentrlaen Strandbjörket, Vaxjo
  - Capio vårdcentralen Hovshaga, Vaxjo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tell D, Tyrstrup M, Edlund C, Rystedt K, Skoog Stahlgren G, Sundvall PD, Hedin K. Clinical course of pharyngotonsillitis with group A streptococcus treated with different penicillin V strategies, divided in groups of Centor Score 3 and 4: a prospective study in primary care. BMC Infect Dis. 2022 Nov 11;22(1):840. doi: 10.1186/s12879-022-07830-4. PMID 36368940
- [Derived] Skoog Stahlgren G, Tyrstrup M, Edlund C, Giske CG, Molstad S, Norman C, Rystedt K, Sundvall PD, Hedin K. Penicillin V four times daily for five days versus three times daily for 10 days in patients with pharyngotonsillitis caused by group A streptococci: randomised controlled, open label, non-inferiority study. BMJ. 2019 Oct 4;367:l5337. doi: 10.1136/bmj.l5337. PMID 31585944